CLINICAL TRIAL: NCT05889468
Title: The Association Between Postpartum Aspirin Use and NT-proBNP Levels as a Marker for Maternal Health Outcomes.
Brief Title: Postpartum ASA and NT-proBNP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00112143
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Treatment Arm vs Placebo Arm
Who Masked: Participant, Investigator
Masking Description: 1:1 fashion to aspirin 81 mg vs identical-appearing placebo to be continued for 6 weeks' postpartum. Patients will receive these medications prior to hospital discharge. Both the patient and provider will be blinded to their assigned group. NT-proBNP levels will be drawn at the 4-6-week postpartum visit. NT-proBNP levels will be compared between groups.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Active Comparator): The treatment group will be provided with a 6-week supply of 81 mg of aspirin prior to discharge from the delivery admission. Patients will be scheduled for a 4-6 week postpartum clinic appointment, which is standard for these patients outside of this proposal.
  Interventions: Drug: Aspirin 81Mg Ec Tab
- Placebo Group (Placebo Comparator): The control group will receive a 6-week supply of placebo medication from the Investigational Pharmacy prior to discharge. The placebo will be identically appearing to the 81 mg aspirin. Patients will be scheduled for a 4-6 week postpartum clinic appointment, which is standard for these patients outside of this proposal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab — Participant may be provided with a 6-week supply of 81 mg of aspirin prior to discharge from the delivery admission.
  Arms: Treatment Group
Drug: Placebo — Participant may be provided with a 6-week supply of placebo to discharge from the delivery admission.
  Arms: Placebo Group

SUMMARY:
This study is a double-blinded randomized-controlled trial in which patients will be randomized to 81 mg of aspirin or placebo to be continued for 6 weeks' postpartum. The purpose of this study is to compare NT-proBNP levels at the 4-6 week postpartum visit between groups. There is currently no data on the maternal health effects associated with continuation of low-dose aspirin in the postpartum period. This study aims to fill a gap in the knowledge regarding the utility of low-dose aspirin following delivery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* English-speaking
* postpartum
* have met USPSTF recommendations for low-dose aspirin use during pregnancy: >1 high risk factor (history of preeclampsia in prior pregnancy, multifetal gestational, chronic hypertension, preexisting diabetes, renal disease, autoimmune disease) or >2 moderate risk factors (nulliparity, obesity, family history of preeclampsia, sociodemographic characteristics, age 35 years or older, or personal history factors) and reported at least 50% compliance with aspirin during pregnancy.

Exclusion Criteria:

* hypersensitivity reaction to aspirin or other salicylates,
* history of gastrointestinal bleeding
* history of gastric or duodenal ulcers
* severe hepatic dysfunction
* bleeding disorders and diathesis
* known cardiac dysfunction with reduced ejection fraction, or are taking or prescribed ACE inhibitors.
* Patients who required ICU level care during their pregnancy will be excluded.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenna Hughes, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting inclusion criteria were approached for enrollment during routine prenatal visits at Duke Perinatal Clinic and on Duke Birthing Center's Labor and Delivery Unit.
Pre-assignment Details: Four participants were consented but did not start the study because they did not deliver within the Duke Hospital System or required Intensive Care Unit (ICU) admission during their delivery hospitalization.
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 55 | 55
Completed | 44 | 51
Not Completed | 11 | 4
Not completed — Lost to Follow-up | 9 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (5.4) | 32.2 (5.9) | 32.0 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 24 | 45
  White | 31 | 26 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 45 | 51 | 96
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: NT-proBNP Levels at 4-6 Weeks Postpartum
Description: The primary outcome for this analysis was NT-proBNP levels collected at the postpartum visit. Patients were reminded of this appointment the day prior to their scheduled follow-up visit. NT-proBNP levels were drawn at the 4-6 week postpartum visit. If patient did not present to their scheduled appointment, attempts were made to contact the patient and reschedule the visit and collect the lab sample for completion of the study.
Time Frame: 4-6 weeks postpartum
Population: Participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
pg/mL | 36.5 [36.0 to 61.0] | 39.5 [36.0 to 74.0]
Statistical Analysis 1: Comparison: Treatment Group vs Placebo Group; This was an intention-to-treat analysis; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test, a non-parametric test, was used since the empirical distribution of data did not follow the normality assumption

2. Secondary Outcome: Number of Participants With Preeclampsia Diagnosis Postpartum
Time Frame: 6 weeks postpartum
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
Participants | 3 | 7
Statistical Analysis 1: Comparison: Treatment Group vs Placebo Group; Intention-to-treat analysis; Test type: Superiority; p = 0.32, Fisher Exact

3. Secondary Outcome: Number of Participants With Eclampsia
Time Frame: 4-6 weeks postpartum
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Hospital Readmission for Blood Pressure Monitoring or Cardiovascular Disease Work-up Indications
Time Frame: 6 weeks postpartum
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
Participants | 3 | 3
Statistical Analysis 1: Comparison: Treatment Group vs Placebo Group; Intention-to-treat analysis; Test type: Superiority; p > 0.99, Fisher Exact

5. Secondary Outcome: Number of Participants Requiring Initiation or Increase in Blood Pressure Medications
Time Frame: 4-6 weeks postpartum
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
Participants | 3 | 4
Statistical Analysis 1: Comparison: Treatment Group vs Placebo Group; Intention-to-treat analysis; Test type: Superiority; p > 0.99, Fisher Exact

6. Secondary Outcome: Number of Participants With Hospital Readmission for Bleeding-related Complications
Time Frame: 4-6 weeks postpartum
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Needing Blood Transfusion(s)
Time Frame: 4-6 weeks postpartum
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 44 | 51
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 4-6 weeks postpartum
Description: Prespecified minor adverse events included GI symptoms or minor bleeding events. Major bleeding, defined by ISTH as 1) fatal bleeding, 2) symptomatic bleeding in a critical organ, or 3) bleeding causing a fall in hemoglobin level of 20 g/l or more or leading to transfusion of 2 or more units of whole blood or red cells, as well as anaphylactic reactions, unexpected hospitalizations, and death were reported as major adverse events.
Arm/Group | Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 5/55 | 6/55
Other Adverse Events (participants affected / at risk) | 2/55 | 5/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=55) | Placebo Group (N=55)
Unexpected hospitalization (preeclampsia or cardiovascular-related) (Cardiac disorders) | 3 | 3
Unexpected hospitalization (bleeding related) (Blood and lymphatic system disorders) | 0 | 1
Unexpected hospitalization (infection or wound complication) (Infections and infestations) | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=55) | Placebo Group (N=55)
Gastrointestinal symptoms (Gastrointestinal disorders) | 0 | 1
Postpartum triage visit (Pregnancy, puerperium and perinatal conditions) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05889468/Prot_SAP_000.pdf